CLINICAL TRIAL: NCT02632058
Title: Efficacy of Treatment for Tinnitus Based on Cognitive Behavioural Therapy in an Inpatient Setting: a 10-year Retrospective Outcome Analysis
Brief Title: Efficacy of Treatment for Tinnitus
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Psychiatrische Dienste Graubuenden (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-not defined
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Cognitive Behavioral Therapy

SUMMARY:
Tinnitus is the acoustic perception of sound without any physical source. It is estimated that 15-21% of adults develop a Tinnitus, which can cause serious distress and debilitation in all aspects of daily life of the affected.

There is currently no evidence for a successful treatment of tinnitus. While one treatment approach involves sound-based therapies, e.g. tinnitus retraining therapy. The treatment aspect in our setting involved cognitive behavioural therapy.

DETAILED DESCRIPTION:
Tinnitus is the perception of sound in the ears or head unrelated to an external source [Nondahl 2011]. It is a common condition with a prevalence of 25.3% (approximately 50 million) among adults in the United States and increasing with age, peaking at age 60 - 69 years [Shargorodsky 2012] and above the age of 55 years respectively [Nondahl 2012]. Of individuals with tinnitus, 7.9% (approximately 16 million) experience frequent tinnitus which involves perception at least once daily [Shargorodsky 2012]. Prevalence of tinnitus in adults in Europe is described at a similar level with 21.2% [Hendrickx 2007]. In Switzerland prevalence for tinnitus in individuals over the age of 15 years is 20%; of these 13% report having a current tinnitus and 7% report of having had tinnitus in the past five years. [Bieri 2012]. It has been shown that the 10-year cumulative incidence for tinnitus is 12.7% [Nondahl 2010]. Gender seems to play a role in the predisposition for tinnitus; prevalence for men is 26.1% and for women 24.6% [Shargorodsky 2012], while the incidence for men is 14.8% and for women 11.2% [Nondahl 2010]. There is indication that there is also a gender-related level of affliction related to tinnitus, so that women feel more distress [Seydel 2013] and emotional disturbance than men [Pajor 2012].

It has also been shown for tinnitus to have a familial occurrence; subjects related to a sibling with tinnitus have a 1.7 times higher probability to have tinnitus than subjects from a family without tinnitus. [Hendrickx 2007]. Tinnitus perceived as severe has a prevalence of 1.3% [Nondahl 2012].

Risk factors for developing tinnitus are numerous and include conditions involving auditory function (i.e. hearing impairment, exposure to noise and history of ear surgery, head injury or otosclerosis), cardiovascular-related (i.e. cardiovascular disease, peripheral vascular disease, obesity, current smoking, higher number of packyears smoked and history of heavy alcohol consumption) [Nondahl 2012].

Tinnitus is also known to be associated with various complaints such as sleep disturbances, which are reported to be greater in elderly people [Hebert 2007], although there seems to be no difference between people suffering from insomnia with or without tinnitus, which was measured in a population of 38-62 year olds [Crönlein 2007]. Furthermore, tinnitus severity significantly correlates with depression and anxiety symptoms [Udupi 2013]. In addition, there is a higher incidence of somatoform disorders in individuals with tinnitus [Zirke 2013]. Although the severity of tinnitus is associated with anxiety and depression, a causality cannot be concluded [Zöger 2006].

Concerning treatment of tinnitus, tinnitus masking and tinnitus retraining therapy are two successfully applied methods. While both methods use counseling and acoustic stimulation for intervention, the main objective in tinnitus masking is to use wide-band noise applied through ear-level devices, in order to provide immediate relief from tinnitus [Henry 2006]. Although both methods show remarkable improvement in ameliorating tinnitus, in comparison the effects of tinnitus retraining therapy improve progressively over time [Henry 2006]. The results of tinnitus retraining therapy also sustain over time [Forti 2009] and improve quality of life of those affected [Seydel 2014].

In recent years there have been numerous publications implementing a therapeutic model based on cognitive behavioral therapy with a sound-focused tinnitus retraining therapy, proving its effectiveness and long-term effects [Herraiz 2005, Robinson 2008, Zenner 2012, Cima 2012], with long-term effects persisting 15 years after completion of the therapy-program [Goebbel 2006]. Also, tinnitus retraining therapy carried out as a short-term therapy in an outpatient setting has also showed to be maintained over time [Mazurek 2009]. Apart from its therapeutic effectiveness tinnitus therapy based on cognitive therapy shows an increased cost-effectiveness compared to usual therapy [Maes 2014].

In the tinnitus-clinic in Chur we have been treating patients with a modified tinnitus-retraining program based on cognitive therapy for a decade. Patients are either admitted by their general practitioner, Otolaryngologist or self-admitted. We offer capacity to treat nation-wide patients in an inpatient setting, for a modified tinnitus retraining therapy lasting four to six-weeks, depending on severity of comorbid factors. Up to date, there is no other clinic in Switzerland treating individuals in an inpatient setting to the likes of ours. Admitted patients usually have a long way of suffering with an unsuccessful search for enduring relief. With this study we intend to show an improvement in treatment of tinnitus based upon our model of modified tinnitus retraining therapy. If our therapeutic model is successful, many individuals could benefit from a substantial improvement in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* minimum age of 18,
* existing Tinnitus auris or capitis

Exclusion Criteria:

* Psychosis,
* serious physical illness,
* Organic psychiatric disability (ICD-10 F0x.x),
* diseases classified under ICD-10 F2x.x,
* Lack of capacity,
* current substance abuse (F10.x - F19.x according to ICD-10, F17.x not included),
* insufficient knowledge of German.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients suffering from chronic tinnitus referred to our clinic by their treating physician. There is a remarkable level of suffering from chronic tinnitus in these individuals. The participants received an established routine treatment as part of multimodal treatment at an inpatient psychiatric facility. Clinical experience shows that the applied treatment poses a low risk and demonstrates a great amount of benefit. At admission to our clinic all participants were of age and able to give their consent to treatment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Tinnitus-severity assessed with the Tinnitus-questionnaire (Goebel and Hiller 1998). | 6-8 weeks

SECONDARY OUTCOMES:
Brief Symptom Inventory (BSI, Derogatis 1975) | 6-8 weeks
Beck Depression Inventory (BDI, Beck 1961) | 6-8 weeks
Noise Sensitivity Questionnaire [Nelting 2004] | 6-8 weeks

IPD SHARING:
Plan to Share IPD: No